CLINICAL TRIAL: NCT03648333
Title: Clinical Trial to Assess the Pharmacokinetic Characteristics of Lodivixx Tab. 5/160mg in Healthy Male Subjects
Brief Title: Clinical Trial to Assess the Pharmacokinetic Characteristics of Lodivixx Tab. 5/160mg in Healthy Male Subjects (N=27)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HL-LDV-103
Record Dates: First submitted 2018-08-02; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Healthy Male Subjects
Keywords: amlodipine; valsartan; hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination; Amlodipine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lodivixx tab. 5/160mg (Experimental): S-amlodipine nicotinate (5mg as S-amlodipine), valsartan 160mg
  Interventions: Drug: Lodivixx tab. 5/160mg
- Exforge tab. 10/160mg (Active Comparator): amlodipine besylate (10mg as amlodipine), valsartan 160mg
  Interventions: Drug: Exforge tab. 10/160mg

INTERVENTIONS:
Drug: Exforge tab. 10/160mg
  Other Names: amlodipine besylate; valsartan
  Arms: Exforge tab. 10/160mg
Drug: Lodivixx tab. 5/160mg
  Other Names: S-amlodipine nicotinate; valsartan
  Arms: Lodivixx tab. 5/160mg

SUMMARY:
To assess the pharmacokinetic characteristics of valsartan and S-amlodipine after single oral administration of Exforge tab. 10/160mg, a combination formulation of valsartan and amlodipine as reference drug and Lodivixx tab. 5/160mg, a combination formulation of valsartan and S-amlodipine as test drug in healthy male adults

DETAILED DESCRIPTION:
The purpose of this study is to assess the pharmacokinetic characteristics of valsartan and S-amlodipine after single oral administration of Exforge tab. 10/160mg, a combination formulation of valsartan and amlodipine as reference drug and Lodivixx tab. 5/160mg, a combination formulation of valsartan and S-amlodipine as test drug in healthy male adults. Additionally the safety and tolerability of two drugs will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Years 20-45
* Body weight ≥ 50kg and 18 ≤ BMI ≤ 29kg/m2
* Volunteer for the study and sign to ICF

Exclusion Criteria:

* Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with symptoms of acute disease within 28 days prior to study medication
* Subject with history which affect on the absorption, distribution, metabolism or excretion of drug
* Subject with clinically significant active chronic disease
* Subject with any of the following conditions in laboratory test i. AST(sGOT) or ALT(sGPT) > Upper normal limit × 1.5 ii. Total bilirubin > Upper normal limit × 1.5 iii. renal failure with Creatinine clearance < 50mL/min
* Clinically significant hypotension when screening period (SBP < 100mmHg, DBP < 60mmHg)
* Positive test results for HBs Ab, HCV Ab, Syphilis regain test
* Use of any prescription medication within 14 days prior to study medication
* Use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
* Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
* Subject with known for hypersensitivity reaction to S-amlodipine, amlodipine and valsartan and dihydropyridine derivatives
* Subject who is not able to taking the institutional standard meal
* Subjects with whole blood donation within 60 days, component blood donation within 20 days
* Subjects receiving blood transfusion within 30 days prior to study medication dosing
* Participation in any clinical investigation within 60 days prior to study medication dosing
* Continued excessive use of caffeine (caffeine > five cups/day), severe heavy smoker (cigarette > 10 cigarettes per day) and alcohol (alcohol>30 g/day)
* Subject who has been taken meal which affect on the absorption, distribution, metabolism, excretion of drug, especially grapefruit juice
* Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 28 days prior to study medication dosing
* Continued serum potassium concentration abnormal status (on baseline visit, < 3.5 mEq/L or > 5.5 mEq/L)
* Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator
* Severe renal insufficient subjects (creatinine clearance : less than 10 mL/min)
* Severe hepatic insufficient subjects,billiary cirrhosis, biliary obstruction and cholestasis patient
* Combination with aliskiren in Diabetic patient or moderate to severe renal insufficient subjects (glomerular filtration rate<60 mL/min/1.73m2)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration) | 0 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 3.5 hour, 4 hour, 4.5 hour, 5 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour, 72 hour
AUC(area under curve) | 0 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 3.5 hour, 4 hour, 4.5 hour, 5 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour, 72 hour

SECONDARY OUTCOMES:
Number of participants with adverse events | 0 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 3.5 hour, 4 hour, 4.5 hour, 5 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour, 72 hour

CONTACTS AND LOCATIONS:
Overall Officials: KyoungSook Kim, PhD, Study Chair — Metro Hospital